CLINICAL TRIAL: NCT02893007
Title: A Randomized Controlled Trial of a Brief Family-centered Care Program for Hospitalized Patients With Bipolar Disorder and Their Caregivers
Brief Title: A Brief Family-centered Care Program for Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Head Nurse, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201002004IA
Record Dates: First submitted 2016-08-28; First posted 2016-09-08 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brief family-centered care program (Experimental): The Brief family-centered care (BFCC) program was developed and provided for hospitalized patients with BPD and their family caregivers.The BFCC protocol is outlined as 4 treatment sessions, specific goals, and example questions. Four 90-minute in-depth sessions for each dyad were initially held in a quiet interview room to assess family function, then to provide information about BPD, to support and empower the dyads to change communication styles and resolve conflicts, and to sustain or improve family function in the cognitive, affective, and behavioral domains.
  Interventions: Other: Brief family-centered care (BFCC) program
- treatment-as-usual (TAU) (No Intervention): All patients were given the standard hospital-provided services: psychiatric nursing care, occupational therapy, and pharmacotherapy. All of the family caregivers were only to attend a routine 60-minute family discussion group about violence and suicide prevention without any specific patient-family dyad interview.

INTERVENTIONS:
Other: Brief family-centered care (BFCC) program — The therapist provided the 4-session BFCC program twice a week for each dyad. The core principles treated family as a single unit and provided individually tailored interventions to improve family function through psychoeducation, social and emotional support, and actively raising questions to facilitate constructive awareness and changes. It was initially held to assess family function, then to provide information about BPD, to support and empower the dyads to change communication styles and resolve conflicts, and to sustain or improve family function in the cognitive, affective, and behavioral domains.
  Arms: Brief family-centered care program

SUMMARY:
Family interventions have been emphasized in the treatment of BPD and have benefits for patients' symptoms and health; however, the effects of family interventions on family function and caregivers' health-related outcomes have not been well investigated. This randomized controlled trial with 47 hospitalized patient-with-BPD/family-caregiver dyads at a medical center in northern Taiwan compared the effects of a brief family-centered care (BFCC) program with treatment-as-usual (TAU). The findings support both the feasibility of using the BFCC program for inpatients and its specific benefits for family function. An intensive family intervention during hospitalization has been suggested in psychiatric practice to support patients with BPD and family caregivers.

DETAILED DESCRIPTION:
All of the family caregivers in two groups were invited to attend a routine 60-minute family discussion group about violence and suicide prevention. The TAU group without specific family interview for patient and family caregiver dyad. In the BFCC group, four 90-minute BFCC program sessions were additionally provided twice a week for each hospitalized family dyad. It was hypothesized that family caregivers in the BFCC group could primary increase their family function, and secondary improve perceived health status and reduce caregiver's burdens compared to the TAU. The results showed family caregivers in the BFCC group significant time group interaction effects in overall family function (p=0.03) and subscale-conflict (p=0.04), communication (p=0.01), and problem solving (p=0.04), but there were no significant interaction effects on the caregivers' perceived health status and caregiver's burdens.

ELIGIBILITY:
Inclusion Criteria:

* Patients were enrolled if they met the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) (American Psychiatric Association 1994) criteria for BP-I or BP-II disorder, were able to be interviewed, and had a Hamilton Depression Rating Scale (HDRS) score < 17 and a Young Mania Rating Scale (YMRS) score < 38 (Keck 2004) to prevent adverse effects caused by patients' mood instability.
* Family caregivers who were identified as: (i) significant in the patient's life, (ii) at least 18 years old, (iii) having lived with the patient for at least 6 months, (iv) able to speak and understand Chinese or Taiwanese, and (v) able to answer questionnaires written in Chinese were included.

Exclusion Criteria:

* Patients who had lived alone or lived with their family for less than 6 months, had been concurrently diagnosed with intellectual disability (DSM-5) (American Psychiatric Association 2013), had been newly diagnosed with BPD at this admission, or could not speak Chinese were excluded.
* Caregivers diagnosed with a serious mental illness or intellectual disabilities were excluded.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change of family function assessed by the Chinese-version Family Functioning Scale (FFS) | To assess the change from baseline through study completion, an average of 4 weeks.
  Self-reported, each item is rated using a 5-point Likert scale, and 11 negative items are reverse-scored. Higher scores indicate better family function.

SECONDARY OUTCOMES:
Change of caregivers' perceived health status assessed by the Chinese Health Questionnaire (CHQ)-12 | All were assessed the change from baseline through study completion, an average of 4 weeks.
  It contains 12 items in four dimensions: physiological and somatic, anxiety and worry, depression and poor relationships, and sleep problems. Each item is rated using a 4-point Likert scale (0-3). Total scores < 3 indicated normal psychological health, and total scores > 3 indicated worsening symptoms and that the patient was at risk for mental problems. Higher scores indicated worsening conditions.
Change of caregivers' burden assessed by the the Chinese-version Caregiver Burden Inventory (CBI) | All were assessed the change from baseline through study completion, an average of 4 weeks.
  The CBI contains 24 items in 5 dimensions: physiological, social, emotional, time, and development. Each item is rated using a 5-point Likert scale (0-4); total scores range from 0 to 96. Higher scores mean greater caregiver burdens.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Ju Lee, MS, Principal Investigator — Head Nurse, Department of Nursing, Taipei Veterans General Hospital, Taipei, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No